CLINICAL TRIAL: NCT03404089
Title: Bedside Therapeutic Monitoring of β-Lactam Levels in Newborns, Children and Adolescents Admitted to Intensive Care: Study of a Pharmacokinetics Monitoring Method.
Brief Title: Bedside Therapeutic Monitoring of β-Lactam Levels in Newborns, Children and Adolescents Admitted to Intensive Care.
Acronym: MON4STRAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient inclusions
Sponsor: University Hospital, Lille (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015_78; 2016-A01407-44 (Other: ID-RCB number, ANSM); HEALTH.2013.2.3.1-2 (Other: FP7-HEALTH-2013-INNOVATION-1)
Record Dates: First submitted 2017-11-28; First posted 2018-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Intensive Care Unit Syndrome
Keywords: device drug monitoring; β-lactam antibiotic; health care-associated infection; MON4STRAT
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pharmacokinetic device (Experimental): MON4STRAT system
  Interventions: Device: pharmacokinetic device

INTERVENTIONS:
Device: pharmacokinetic device — MON4STRAT system: bed-side pharmacokinetic device for drug concentration measurement
Device: pharmacokinetic device — High performance liquid chromatography, (HPLC), the reference methods HLPC tandem mass spectrometry or Ultraviolet are using

SUMMARY:
This study evaluate the capacity of the MON4STRAT device for drug monitoring of β- lactam antibiotic concentrations in newborns, children, and adolescents admitted in intensive care units with a health care-associated infection.

ELIGIBILITY:
Inclusion Criteria:

* Age younger than 18 years
* Newborns (preterm or not) in neonatal intensive care
* Infants, children, and adolescents in pediatric intensive care
* Clinically suspected or microbiologically proven sepsis that might be associated with ventilator-associated pneumonia or otherwise associated with health care
* Need for antibiotic treatment by piperacillin-tazobactam, ceftazidime, or meropenem of intermittent administration
* Informed consent form signed by parents/guardian
* Informed consent form signed by patients old enough to understand.

Exclusion Criteria:

* Process for active limitation of treatment underway
* Suspected or known hypersensitivity to studied beta-lactams
* Renal failure, defined as serum creatinine > 1.5 mg/dl or urine production < 0.3 ml/kg for 24 h or anuria for 12 h.
* Co-administration of two β-lactam antibiotics
* Cystic fibrosis
* No national health insurance coverage in French center
* Family unable to understand study-related information due to language or other communication issues
* No consent obtained

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Correlation between the β-lactam dosage measured by the MON4STRAT method and the β-lactam dosage measured by the HPLC-MS-MS (the reference method). | at 3 days

SECONDARY OUTCOMES:
User's questionnaire | at 3 days
  The feasibility of the MON4STRAT method will be evaluated by a questionnaire to be completed by the users of the method, that is, the nurses caring for these patients.
Minimum concentration of beta-lactams antibiotics | before antibiotic infusion at day 3 and 2/3 hours after the end of antibiotic infusion
  Pharmacokinetic of beta-lactams antibiotics
Maximum concentration (CMax) of beta-lactams antibiotics | before antibiotic infusion at day 3 and 2/3 hours after the end of antibiotic infusion
  Pharmacokinetic of beta-lactams antibiotics
Clearance (Cl) of beta-lactams antibiotics | before antibiotic infusion at day 3 and 2/3 hours after the end of antibiotic infusion
  Pharmacokinetic of beta-lactams antibiotics
Volume of distribution of beta-lactams antibiotics | before antibiotic infusion at day 3 and 2/3 hours after the end of antibiotic infusion
  Pharmacokinetic of beta-lactams antibiotics
Half-life (t1/2) of beta-lactams antibiotics | before antibiotic infusion at day 3 and 2/3 hours after the end of antibiotic infusion
  Pharmacokinetic of beta-lactams antibiotics
Assessment of the course of infection of children who had a β-lactam assay (by the reference method) at the usual levels and those who appeared to receiving inadequate β-lactam doses. | at 17 days
  Antimicrobial doses, serum concentration of β- lactams and minimum inhibitory concentration of microorganisms, if available, will be used to assess the potential usefulness of this bedside method

CONTACTS AND LOCATIONS:
Overall Officials: François DUBOS, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France